CLINICAL TRIAL: NCT02248740
Title: Radiofrequency Ablation vs. Laser Ablation of the Incompetent Small Saphenous Vein: A Prospective Randomized Trial
Brief Title: Radiofrequency Ablation vs. Laser Ablation of the Incompetent Small Saphenous Vein
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM11844
Record Dates: First submitted 2014-09-02; First posted 2014-09-25 (Estimated); Results first posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-09

CONDITIONS: Chronic Venous Insufficiency
Keywords: chronic venous insufficiency; varicose vein; small saphenous vein
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency Ablation (Active Comparator): Device: ClosureFast radiofrequency catheter (VNUS Medical Technologies Inc, San Jose, CA).
  Patients will have the intervention, ablation of the incompetent small saphenous vein, using this device.
  Interventions: Procedure: Ablation of the incompetent small saphenous vein
- Laser Ablation (Active Comparator): Device: EVLT 980nm diode laser system (Angiodynamics, Queensbury, NY).
  Patients will have the intervention, ablation of the incompetent small saphenous vein, using this device.
  Interventions: Procedure: Ablation of the incompetent small saphenous vein

INTERVENTIONS:
Procedure: Ablation of the incompetent small saphenous vein — For each patient, the Small Saphenous Vein (SSV) will be accessed from the midcalf. After liberal use of tumescent anesthesia, ablation of the incompetent small saphenous vein will be performed. Half the patients will have this procedure performed using the Laser Ablation device and half will be performed using the Radiofrequency Ablation device. They will be randomly assigned to treatment.

SUMMARY:
The aim of this study is to perform a randomized, prospective trial comparing the two current methods of treatment for chronic venous insufficiency related to the Small Saphenous Vein (SSV) to evaluate complications and outcomes for each method, and ultimately, to see if one is superior to the other.

DETAILED DESCRIPTION:
Chronic venous insufficiency (CVI) is estimated to affect 25 million Americans. This condition leads to varicose veins, aching, fatigue, swelling, ulcerations, and bleeding in the lower extremities. The second most common cause is a refluxing or incompetent Small Saphenous Vein (SSV). This condition results in pooling of deoxygenated blood in the lower extremities rather than successful transport of the blood back to the heart and lungs. The historical treatment has been to surgically remove or 'strip' the SSV so that blood is rerouted through the healthier deep veins. A less invasive treatment option, Endovenous Thermal Ablation, has emerged over the last decade and has virtually replaced stripping. This involves advancing a catheter under ultrasound guidance through the SSV and then advancing a laser fiber or radiofrequency probe through the catheter. These devices then produce the energy to destroy the vein as the catheters are slowly pulled back. While both radiofrequency ablation and laser ablation are accepted treatments, neither technology has been definitively proved to have fewer complications or superior results. This is in part because very few practices have the ability to make a head to head comparison between the two technologies and must choose one or the other secondary to financial constraints. The aim of this study is to perform a randomized prospective trial comparing the two modalities so that more definitive information to evaluate complications and outcome can be obtained and then recommendations on which, if either, technology is superior can be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic chronic venous insufficiency.
* Patients in whom endovenous thermal ablation is clinically indicated.
* Have previously undergone at least 6 weeks of conservative treatment with compression stockings (unless they have venous ulcers, recurrent phlebitis, or bleeding varices).
* Have symptoms secondary to Small Saphenous Vein insufficiency defined as reverse flow in the saphenous vein >0.5 seconds after calf compression or while standing.

Exclusion Criteria:

* Have previously undergone surgery, EVTA, or phlebectomy in that extremity (exclusive of spider vein injections or other cosmetic surface procedures).
* Have a history of Deep Venous Thrombosis (DVT).
* Have a history of hypercoaguability disorder.
* Are pregnant or breastfeeding.
* Are nonambulatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Sydnor, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiofrequency Ablation: Device: ClosureFast radiofrequency catheter (VNUS Medical Technologies Inc, San Jose, CA).
  Patients will have the intervention, ablation of the incompetent small saphenous vein, using this device.
  Ablation of the incompetent small saphenous vein: For each patient, the Small Saphenous Vein (SSV) will be accessed from the midcalf. After liberal use of tumescent anesthesia, ablation of the incompetent small saphenous vein will be performed. Half the patients will have this procedure performed using the Laser Ablation device and half will be performed using the Radiofrequency Ablation device. They will be randomly assigned to treatment.
- Laser Ablation: Device: EVLT 980nm diode laser system (Angiodynamics, Queensbury, NY).
  Patients will have the intervention, ablation of the incompetent small saphenous vein, using this device.
  Ablation of the incompetent small saphenous vein: For each patient, the Small Saphenous Vein (SSV) will be accessed from the midcalf. After liberal use of tumescent anesthesia, ablation of the incompetent small saphenous vein will be performed. Half the patients will have this procedure performed using the Laser Ablation device and half will be performed using the Radiofrequency Ablation device. They will be randomly assigned to treatment.
Period: Overall Study
Arm/Group | Radiofrequency Ablation | Laser Ablation
Started | 18 | 18
Completed | 0 | 0
Not Completed | 18 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiofrequency Ablation | Laser Ablation | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Clinical Symptoms of an Incompetent Small Saphenous Vein After Treatment.
Time Frame: At 10 years after treatment.
Population: No study data was collected prior to study termination.
Arm/Group | Radiofrequency Ablation | Laser Ablation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence Rate of Acute Complications
Time Frame: 1 and 6 weeks post intervention.
Population: No study data was collected prior to study termination.
Arm/Group | Radiofrequency Ablation | Laser Ablation
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Incidence of Pain and Bruising
Description: Measurement of pain will be performed by patient solicitation of pain rating on a scale of 0 to 10.
  Bruising will be measured on a scale of 0-10, determined by a consensus of all study investigators.
Time Frame: During Intervention and post procedure recovery period in clinic, an expected average of 2 hours.
Population: No study data was collected prior to study termination.
Arm/Group | Radiofrequency Ablation | Laser Ablation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Radiofrequency Ablation | Laser Ablation
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT02248740/Prot_SAP_000.pdf